CLINICAL TRIAL: NCT06561763
Title: TPC Versus GP Induced Chemotherapy Combined With Nimotuzumab and Toripalimab in the Treatment of Localized Advanced Nasopharyngeal Carcinoma:Multi Center, Open Label, Randomized Controlled, Non Inferiority Design, Phase III Clinical Study
Brief Title: TPC VS. GP Induced Chemotherapy Combined With Nimotuzumab and Toripalimab in the Treatment of Locally Advanced Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, XIANG YANQUN, chief physician, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYSKY-2024-568-02
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: High Risk Locally Advanced Nasopharyngeal Carcinoma
MeSH Terms: interventions — nimotuzumab; Capecitabine; Gemcitabine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPC+Triprolizumab+Nimotuzumab (Experimental)
  Interventions: Drug: Nimotuzumab,Toripalimab，Cisplatin, albumin paclitaxel, capecitabine
- GP+Triprolizumab+Nimotuzumab (Active Comparator)
  Interventions: Drug: Nimotuzumab,Toripalimab，Cisplatin, Gemcitabine

INTERVENTIONS:
Drug: Nimotuzumab,Toripalimab，Cisplatin, albumin paclitaxel, capecitabine — Albumin paclitaxel 200g/m2, intravenous drip administration, d1; Cisplatin 60 mg/m2， Intravenous , d1; Capecitabine, 1000mg/m2, orally administered D1-14； Triprolizumab injection 240mg, intravenous D1; Nivolumab 400mg, intravenous D1; Q3W 1 cycle, 3 cycles Period, 3 weeks in total
  Arms: TPC+Triprolizumab+Nimotuzumab
Drug: Nimotuzumab,Toripalimab，Cisplatin, Gemcitabine — Cisplatin 80 mg/m2， Intravenous drip administration, d1; Gemcitabine, 1000mg/m2,Intravenous ，D1,D8； Triprolizumab injection 240mg, intravenous ； Nivolumab 400mg, intravenous； Q3W 1 cycle, 3 cycles
  Arms: GP+Triprolizumab+Nimotuzumab

SUMMARY:
We expect to conduct a clinical trial in high-risk locally advanced nasopharyngeal carcinoma patients to explore the efficacy and safety of sequential radical radiotherapy treatment after induction chemotherapy (TPC vs. GP) with combination therapy of nivolumab and triprolizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18-65 years old;
2. Diagnosed with nasopharyngeal carcinoma through histopathology or cytology;
3. Advanced nasopharyngeal carcinoma, AJCC 8th standard stage III-IVA, excluding T3-4N0/T3N1;
4. ECOG score is 0-1;
5. Sufficient organ or bone marrow function:
6. Sign a written informed consent form

Exclusion Criteria:

1. Diagnosed with other malignant tumors within 5 years prior to the first administration, excluding curative basal cell carcinoma, squamous cell carcinoma, and/or excised carcinoma in situ.
2. Symptomatic congestive heart failure, with echocardiogram indicating a left ventricular ejection fraction (LVEF)<50%.
3. Individuals infected with acute or chronic active hepatitis B or C, with hepatitis B virus (HBV) DNA>2000IU/ml or 10^4 copies/ml; Hepatitis C virus (HCV) RNA>10^3 copies/ml; Hepatitis B surface antigen (HbsAg) and anti HCV antibody were positive at the same time. After nucleotide antiviral treatment, if the score is lower than the above standard, it can be included in the group.
4. Past and current history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, drug-related pneumonia, severe impairment of lung function, and other lung diseases.
5. Individuals with active pulmonary tuberculosis (TB) who are currently receiving anti tuberculosis treatment or have received anti tuberculosis treatment within one year prior to their first dose.
6. Human immunodeficiency virus (HIV) infected individuals (HIV 1/2 antibody positive), known syphilis infections requiring treatment.
7. Severe infections that are active or poorly controlled clinically. Within 4 weeks prior to the first administration, there was a severe infection, including but not limited to hospitalization due to infection, bacteremia, or complications of severe pneumonia.
8. An active autoimmune disease requiring systemic treatment (such as the use of disease relieving drugs, corticosteroids, or immunosuppressants) has occurred within 2 years prior to the first administration. Allow the use of alternative therapies such as thyroid hormone, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency. Known history of primary immunodeficiency. Only patients with positive autoimmune antibodies need to confirm the presence of autoimmune diseases based on the researcher's judgment.
9. Pregnant or lactating female patients.
10. Has received radiotherapy, chemotherapy, or surgical treatment for nasopharyngeal and neck lesions (excluding biopsy).
11. History of allergies to the drugs and their components used in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2028-08-20 (Estimated); Study Completion 2031-08-20 (Estimated)

PRIMARY OUTCOMES:
3-year event free survival | 3 years

SECONDARY OUTCOMES:
adverse effects | 3 years
  chemotherapy side effectst
3-year overall survival | 3 years
3-year distant disease free survival | 3 years
3-year local recurrence free survival rate | 3 years

IPD SHARING:
Plan to Share IPD: No